CLINICAL TRIAL: NCT06371443
Title: The Effects of Sucking and Swallowing Exercises on the Transition Process to Oral Feeding in Premature İnfants
Brief Title: Suction and Swalloing Exercises for Premature Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ayselkokcudogan
Record Dates: First submitted 2022-08-19; First posted 2024-04-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Premature Infant
Keywords: Oral feeding; sucking-swallowing exercises; premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 41 premature infants in the experimental group
  Interventions: Behavioral: Sucking and swallowing exercises
- control group (No Intervention): 41 premature infants in the control group

INTERVENTIONS:
Behavioral: Sucking and swallowing exercises — Sucking-swallowing exercises were applied to premature infants in the experimental group (n=41) for 14 days, once a day, 12 minutes before feeding.
  Arms: experimental group

SUMMARY:
Underdeveloped oral structures of preterm infants cause feeding problems. Therefore, the development of sucking reflexes of premature babies should be supported.

This study aimed to investigate the effect of suck-swallow training on the transition to oral feeding in premature infants.

The study was conducted as a randomized controlled experimental trial in the NICU of a public hospital in Istanbul. The study sample consisted of 82 premature infants. Of these infants, 41 were assigned to the experimental group and 41 to the control group. Study data were collected using the investigator-developed Premature Infant Data Collection Form and Early Feeding Skills Assessment Tool. Throughout the study, preterm infants in the experimental group (n=41) were given suck-swallow exercises for 12 minutes once a day before feeding for 14 days. SPSS21 was used to analyze the data.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled experimental study to evaluate the effect of sucking and swallowing training on the transition to oral feeding in premature infants. The study sought to answer the question, "Do suckling and swallowing exercises have an effect on the transition to oral feeding?". The study was carried out between December 2021 and June 2022 at the neonatal intensive care unit of a public hospital in Istanbul. The study sample consisted of infants who were admitted to the neonatal intensive care unit of a public hospital in Istanbul, who met the inclusion criteria, and whose parents consented to the study. A power analysis was performed to determine the number of subjects to be included in the study. The power of the test was calculated using the G*Power 3.1 program. Infants enrolled in the study were randomized in order of arrival to avoid bias. The randomization table was generated by "https://www.calculatorsoup.com" as follows.

Data were collected using the Premature Infant Data Collection Form and the Early Feeding Skills Assessment Tool.

The premature infant data collection form developed by the investigators consists of 2 parts. The first part contains descriptive information about the parents (gender, age, education level, number of children, social security). The second part contains descriptive details of the infant (sex, mode of delivery, Apgar score, week of birth, postmenstrual week at enrollment, birth weight, weight at enrollment, head circumference-height at birth, phototherapy status within the last 24 hours, oxygen support status).

Application in the experimental group: Informed consent was obtained from the parents of the infants in the experimental group who had low suckling success and met the inclusion criteria. After completing the premature infant data collection form, the investigator assessed the infant's sucking activity. Infants with no suck reflex were included in the study group. The oral motor stimulation exercises developed by Fucile and applied to the infants in the experimental group who needed suckling and swallowing exercises were evaluated according to the Early Feeding Skills measurement tool. The investigator performed the exercises on the infants once a day for 12 minutes before feeding for 14 days. After 14 days, the infants were assessed again using the EFS scale.

Application in the control group: First, informed consent was obtained from the parents of the infants in the control group who met the inclusion criteria. After completing the premature infant data collection form, the infant's sucking activity was assessed. Infants who did not show a suck reflex were included in the study group, and the infants were evaluated using the Early Feeding Skills (EFS) measurement tool at baseline and at 14 days.

The data collected in the study were analyzed using SPSS (Statistical Package for Social Sciences) 22.0 for Windows software. Numbers, percentages, means, and standard deviations were used as descriptive statistical methods to analyze the data. Kurtosis and skewness values were examined using chi-square and t-tests to determine whether the study variables were normally distributed.

The study was conducted after obtaining the necessary permissions from XXXXXXXX Non-Interventional Clinical Research Ethics Committee (decision number: 1054, date: 26.10.2021) and the hospital where the study was to be conducted, as well as the informed consent of the parents who consented their children to participate in the study. Infants enrolled in the study were not exposed to practices or procedures that would violate patient rights, that parents would consider inappropriate, or that would adversely affect the patient.

ELIGIBILITY:
Inclusion criteria

* Premature babies with an updated gestational week of 34 weeks
* Premature babies born at 34-37 weeks of gestation
* Premature babies with stable vital signs
* Premature babies with underdeveloped sucking activity

Exclusion criteria

* intubated babies
* Babies with multiple anomalies
* Babies with asphyxia
* Infants with unstable vital signs

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The early feeding skills assessment tool (EFS) | December 2021 and June 2022
  This scale is a reliable tool that assesses skills that contribute to safe and successful oral feeding of preterm infants in 5 sub-dimensions. Sub-dimensions include respiratory regulation, oral motor function, swallowing coordination, feeding participation, and physiological stability.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Arslan, Principal Investigator — Medipol University; Aysel Kokcu Dogan, Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gokdemir E, Dogan AK. The Effect of Suckling and Swallowing Exercises During the Transition to Oral Feeding in Premature Infants: Randomized Controlled Study. Niger J Clin Pract. 2025 Jun 1;28(6):708-715. doi: 10.4103/njcp.njcp_41_25. Epub 2025 Jun 25. PMID 40556083